CLINICAL TRIAL: NCT05970185
Title: Fuling Zhou, Head, Division of Hematology; Professor of Hematology; Doctoral Advisor, Zhongnan Hospital
Brief Title: The Value of Peripheral Blood CD34+ Cell Dynamics Monitoring in Autologous Hematopoietic Stem Cell Transplant Mobilization
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Fuling Zhou, Head, Division of Hematology; Professor of Hematology; Doctoral advisor, Zhongnan Hospital, Zhongnan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07
Record Dates: First submitted 2023-07-12; First posted 2023-08-01 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Granulocyte Colony-Stimulating Factor
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG-rhG-CSF (Experimental): Subcutaneous injection of polyethylene glycolized recombinant human granulocyte-stimulating factor injection 6mg bid in the experimental group the day after the end of chemotherapy
  Interventions: Drug: PEG-rhG-CSF
- G-CSF (Active Comparator): G-CSF 5ug/kg/d from day 5 after the end of chemotherapy until the end of collection
  Interventions: Drug: G-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — Subcutaneous injection of polyethylene glycolized recombinant human granulocyte-stimulating factor injection 6mg bid in the experimental group the day after the end of chemotherapy
  Arms: PEG-rhG-CSF
Drug: G-CSF — G-CSF 5ug/kg/d from day 5 after the end of chemotherapy until the end of collection
  Arms: G-CSF

SUMMARY:
The aim of this study was to evaluate the difference in the accuracy of CD34+ cell detection by immunomagnetic bead method and flow cytometry in patients with hematologic malignancies pre-treated with stem cell transplantation after mobilization, and the results were compared simultaneously in the groups applying different mobilization protocols.

DETAILED DESCRIPTION:
Treatment programs The mobilization protocol is.

1. etoposide 0.1 grams per square meter qd d1-3
2. algocytidine 0.5 grams per square meter q12h d1-3
3. whitening injection (subcutaneous injection of polyethylene glycolized recombinant human granulocyte-stimulating factor injection 6mg bid in the experimental group on the second day after chemotherapy, and G-CSF 5ug/kg/d in the control group from the fifth day after chemotherapy until the end of collection).

In both groups, routine blood tests were performed daily, and the percentage of CD34+ cells in peripheral blood was monitored from the time leukocytes started to rise after the nadir by immunomagnetic bead assay and flow cytometry, and collection was initiated if the percentage of CD34+ was >0.1% and peripheral blood leukocytes were >3.5×109/L.

Collection was stopped when the CD34+ cell count was >5×106/kg, and no more than three attempts were made. Collection was considered a failure when CD34+ cells collected in any of the three attempts did not reach 2×106/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Malignant lymphoma diagnosed by histology and/or cytology; expected survival > 3 months.
2. Patients evaluated for disease in complete or partial remission.
3. Normal bone marrow hematopoietic function; no significant cardiac or pulmonary dysfunction.
4. Liver function and biochemical tests need to meet the following criteria. ALT and AST ≤ 1.5×ULN. TBIL≤1.5×ULN. Blood creatinine ≤ 1.5 × ULN.
5. PS score of 0-2.
6. Age ≥ 18.
7. Women of childbearing potential must have had a pregnancy test (serum or urine) within 7 days prior to enrollment with a negative result and be willing to use an appropriate method of contraception for the duration of the trial.

Subjects voluntarily enrolled in the study, signed an informed consent form, were compliant and cooperated with the follow-up.

Exclusion Criteria:

1. Pregnant or lactating women.
2. having other hematological disorders affecting the hematopoietic function of the bone marrow
3. those with acute or active infections who have received systemic anti-infective therapy within 72h
4. who are allergic to the study drug or other G-CSF products, or to biological agents expressed by E. coli
5. Those who, in the judgment of the investigator, have a serious concomitant disease that jeopardizes patient safety or interferes with the patient's ability to complete the study
6. Other conditions that, in the judgment of the investigator, are not suitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Total CD34+ cell yield (106/kg) | through study completion, an average of 1 year
  Total CD34+ cell yield (106/kg)

SECONDARY OUTCOMES:
Accuracy differences between immunomagnetic bead assays and flow cytometry assays | through study completion, an average of 1 year
  Differences in the accuracy of immunomagnetic bead assay and flow cytometry in the detection of CD34+ cells after mobilization in lymphoma patients prepped for stem cell transplantation
Height | One day before chemotherapy
  height in meters
Weight | One day before chemotherapy
  Weight in kg
Vital signs and physical examination | One day before chemotherapy
  Exclude unrelated organic disease by imaging studies
ECOG score (d1 pre-chemotherapy) | One day before chemotherapy
  The ECOG scoring standard (Eastern Cooperative Oncology Group) is an index to understand the patient's general health status and tolerance to treatment from the patient's physical strength. The patient's activity status is divided into 6 grades from 0 to 5, with higher scores indicating worse outcomes.
Blood routine | Blood routine was tested daily, an average of 1 year
  Blood routine: Blood routine was tested daily, and peripheral blood CD34+ cell percentage was monitored from the time leukocytes started to rise after the nadir by immunomagnetic bead assay and flow cytometry, and collection was initiated if CD34+ percentage was >0.1% and peripheral blood leukocytes were >3.5×109/L.
Adverse event record | through study completion, an average of 1 year
  Adverse event record: record any adverse events that occurred during the drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Fuling Zhou, Study Director — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No